CLINICAL TRIAL: NCT01092312
Title: Study on the Signature Personalised Patient Care System With the Vanguard Knee System
Brief Title: Signature Personalised Patient Care System With the Vanguard Knee System Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No difference in outcome between the two groups
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBMET.CR.G4
Record Dates: First submitted 2010-03-07; First posted 2010-03-24 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: knee; arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Signature Knee Guide (Experimental): Vanguard Knee System with Signature Knee Guide
  Interventions: Procedure: Vanguard Knee System with Signature Knee Guide
- Conventional Approach (Active Comparator): Vanguard Complete Knee System with Conventional Approach
  Interventions: Procedure: Vanguard Knee System with conventional Instruments

INTERVENTIONS:
Procedure: Vanguard Knee System with Signature Knee Guide — Use of Signature Knee Guide
  Arms: Signature Knee Guide
Procedure: Vanguard Knee System with conventional Instruments — Vanguard Knee System with conventional Instruments
  Arms: Conventional Approach

SUMMARY:
The purpose of this study is to determine whether the percentage cases which have ideal mechanical axial alignment using the Vanguard total Knee implant with the Signature cutting blocks is higher than those without the use of Signature when measured immediately post-operatively.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the percentage cases which have ideal mechanical axial alignment using the Vanguard total Knee implant with the Signature cutting blocks is higher than those without the use of Signature when measured immediately post-operatively. Other outcomes will include knee assessments and patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more of the knee compartments are involved
* correction of varus, valgus or posttraumatic deformity
* correction or revision of unsuccessful osteotomy (wedge cut from bone to improve alignment), or arthrodesis (fusion)
* need to obtain pain relief and improve function
* ability and willingness to follow instructions, including control of weight and activity level.
* a good nutritional state
* must have reached full skeletal maturity
* able and willing to undergo an MRI scan

Exclusion Criteria:

* infection
* sepsis
* osteomyelitis
* failure of a previous joint replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Mechanical Axial Alignment | Prior to Discharge: 0-2 weeks
  Femoral and tibial component alignment, femoral and tibial rotational alignment, tibial posterior slope

SECONDARY OUTCOMES:
Clinical Outcome | 6 months, 1 year
  American Knee Society Score, Oxford Knee Score

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Morrison, MBChB, Principal Investigator — The Queen Elizabeth Hospital
Locations (12):
- Insall Scott Kelly Institute, New York, New York, United States
- Australia (2):
  - Logan Hospital, Brisbane, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
- Austria (2):
  - General Hospital Kreuzschwestern, Grieskirchen, Wels
  - The Orthopaedic Hospital Speising, Vienna
- St Luc General Hospital, Brussels, Belgium
- Aalborg University Hospital, Aalborg, Denmark
- Medipole de Savoie, Chambéry, France
- Amphia Ziekenhuis Breda, Breda, Netherlands
- Torres Verdras Hospital, Torres Vedras, Lisbon District, Portugal
- Danderyd Hospital, Stockholm, Sweden
- Addenbrooke's Hospital, Cambridge, United Kingdom